CLINICAL TRIAL: NCT03548389
Title: The Effect of Mother and Newborn Early Skin-to-skin Contact on Initiation of Breastfeeding, Newborn Temperature and Duration of Third Stage of Labor
Brief Title: The Effect of Early Skin-to-skin Contact on Initiation of Breastfeeding, Newborn Temperature and Duration of Third Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Kolsoom Safari, Investigator, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2
Record Dates: First submitted 2018-05-23; First posted 2018-06-07 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother and newborn skin to skin contact (Experimental): By assistance of the researcher, intervention infants were placed undressed in a prone position against their mothers' bare chest between breasts immediately after birth and before placental delivery and suturing of tears or episiotomy. The Apgar score was determined, the infant's nose and mouth were suctioned while on the mother's chest, it was well dried, and both mother and infant were covered with a pre-warmed blanket. To prevent heat loss, the infant's head was covered with a dry cap that was replaced when it became damp. Dressing and measuring of the infant were postponed to an hour after the delivery by registered midwife.
  Interventions: Other: Skin to skin contact
- Conventional care (No Intervention): In the routine care group, the infant was delivered from the mother by a midwife, wrapped in blankets, taken to be routinely cared under a warmer, and then dried quickly. Afterwards, the Apgar score was determined immediately after the umbilical cord was cut. The infants were provided with all routine care by the midwife working in the delivery room. After the infants were weighed, dressed, and measured, they were handed to their mothers who were encouraged to begin breastfeeding.

INTERVENTIONS:
Other: Skin to skin contact — By assistance of the researcher, intervention infants were placed undressed in a prone position against their mothers' bare chest between breasts immediately after birth and before placental delivery and suturing of tears or episiotomy. The Apgar score was determined, the infant's nose and mouth were suctioned while on the mother's chest, it was well dried, and both mother and infant were covered with a pre-warmed blanket. To prevent heat loss, the infant's head was covered with a dry cap that was replaced when it became damp. Dressing and measuring of the infant were postponed to an hour after the delivery by registered midwife.
  Arms: Mother and newborn skin to skin contact

SUMMARY:
Background: Keeping mother and newborn skin-to-skin contact (SSC) after birth brings about numerous protective effects; however, it is an intervention that is underutilized in Iraq where a globally considerable rate of maternal and child death has been reported. The present study was carried out in order to assess the effects of mother and newborn skin-to-skin contact on initiation of breastfeeding, newborn temperature, and duration of the third stage of labor.

Methods: A quasi-experimental study was conducted on 108 healthy women and their neonates (56 in the intervention group with mother and newborn skin-to-skin contact and 52 in the control group that were provided with routine postpartum care) at maternity teaching hospital of Erbil, Iraq from February to May, 2017. The required data were collected using four instruments. The first instrument was a structured interview to elicit socio-demographic and obstetric characteristics from the participants. The second instrument was a form that was used to assess the duration of the third stage of labor in mothers. The third instrument was a form to record the newborns' axillary temperature. The fourth instrument was the LATCH scale that was employed to assess the success of the first breastfeed.Descriptive relationships between demographic variables and type of care provided for mothers and newborns after birth were explored using means and SD for continuous variables, whilst categorical variables were described using proportions. The relationship between SSC and time to initiate breastfeeding, duration of third stage of labour, success of breastfeeding, newborn hypothermia, and temperature of the newborn 30 minutes after birth were examined using T test and Chi square. In logistic regression model, the effect of SSC and conventional care on outcomes of the study was analysed by adjusting of potential confounders like mother's age, education level, occupation, number of parity, and newborn gender.

ELIGIBILITY:
Inclusion Criteria:

* healthy women with term singleton pregnancy

Exclusion Criteria:

* low APGAR score in Newborn

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Early initiation of breastfeeding | Immediately After birth
  Time to initiate breastfeeding
Third stage of labour | birth
  Duration of third stage of labour
Newborn temperature | 30 minutes after birth
  Newborn temperature 30 minutes after birth
Success of first breastfeeding | Immediately after birth
  Success of first breastfeeding assessed by LATCH scale

CONTACTS AND LOCATIONS:
Locations (1):
- Kolsoom Safari, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
I would make IPD available if any researcher required them , since I I save my participants information by coding.

REFERENCES:
- [Derived] Safari K, Saeed AA, Hasan SS, Moghaddam-Banaem L. The effect of mother and newborn early skin-to-skin contact on initiation of breastfeeding, newborn temperature and duration of third stage of labor. Int Breastfeed J. 2018 Jul 16;13:32. doi: 10.1186/s13006-018-0174-9. eCollection 2018. PMID 30026787